CLINICAL TRIAL: NCT00468507
Title: The Anti-inflammatory Effects of High-fat Nutrition; Towards a Clinical Application
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: J.W.M. Greve, MD, PhD, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 067030
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Trauma
Keywords: CCK release
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: nutritional intervention with Respifor and Diasip — Four nutritional interventions on four separate days per test person

SUMMARY:
Patients undergoing major surgery, trauma and burns are prone to develop an exacerbated inflammatory response, which is potentially lethal to the individual. Recently our group demonstrated that administration of high fat feeding prior to hemorrhagic shock attenuates severe inflammation, gut barrier loss and hepatic damage. High fat feeding releases cholecystokinin in the gut, which stimulates the autonomous nervous system and subsequently activates the efferent vagus nerve. The activated efferent fibers inhibit tissue macrophages via binding of acetylcholine to the alpha7-nicotinergic receptor.

In this study the cholecystokinin release in healthy volunteers is monitored in response to low fat and high fat food products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* 45 > age <55

Exclusion Criteria:

* Gastrointestinal diseases
* Inflammatory conditions

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
CCK-release | two hours

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Greve, professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Maastricht, Maastricht, Limburg, Netherlands